CLINICAL TRIAL: NCT01735552
Title: Transfusion-related Inflammatory Cytokine and Neutrophil Extracellular Trap Quantification in Neonates.
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 51050
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Anemia of Prematurity; Necrotizing Enterocolitis
Keywords: gut reperfusion injury; blood transfusions; premature infants; anemia; regional oxygen saturations; necrotizing enterocolitis; mesenteric oxygenation
MeSH Terms: conditions — Anemia; Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants requiring PRBCs: Premature infants who require PRBCs for anemia that is not related to sepsis, surgery, NEC or immunologic abnormalities.

SUMMARY:
Despite many advances in neonatal care, necrotizing enterocolitis (NEC) remains a leading cause of morbidity and mortality among premature infants. NEC is the most common life-threatening gastrointestinal emergency encountered in the neonatal intensive care unit, affecting between 3.8% and 13% of very low birthweight (VLBW) infants (1-3). More recently interest has intensified regarding the possible association between "elective" red blood cell (RBC) transfusions in premature infants and the subsequent development of NEC (4-9). On a physiological basis, a few explanations for transfusion-associated NEC have been proposed: 1) the physiological impact of anemia that can initiate a cascade of events leading to ischemic-hypoxemic mucosal gut injury predisposing to NEC [10]; and 2) increased splanchnic blood flow following RBC transfusion leading to reperfusion injury of gut mucosa.

Aim 1. This study will quantify inflammatory cytokine profiles in anemic infants cared for in the NICU prior to and after transfusion with packed red blood cells (PRBC), as dictated by current clinical guidelines for treatment of anemia, and prospectively assess for clinical signs and symptoms of NEC following each transfusion event.

Aim 2. Polymorphonuclear leukocytes (PMNs) isolated from the pre- and post-transfusion blood samples will be assessed in vitro for neutrophil extracellular traps (NET) formation.

Aim 3. A) To determine whether significant anemia preceding a RBC transfusion is associated with impaired intestinal oxygenation, and whether a RBC transfusion temporarily increases splanchnic oxygenation. We postulate that the CSOR will be low (<0.75) at baseline measurement in infants with hemodynamically significant anemia, and that RBC transfusion will temporarily increase intestinal perfusion in that particular group of babies.

B) To determine whether alterations in mesenteric regional oxygenation saturation(rSO2) can predict the development of NEC in VLBW infants. We hypothesize that overall cerebro-splanchnic oxygenation ratio (CSOR) values will be significantly lower among very low birth weight (VLBW) infants that develop NEC, when compared to CSOR values obtained in infants that do not develop NEC following RBC transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient in NICU at UUMC, PCMC, or IMC
* Gestational age at birth ≤ 32 weeks
* Birth weight ≤ 1500 grams
* Age ≤ 12 weeks of life

Exclusion Criteria:

* Lack of parental consent
* Multiple congenital anomalies

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted into the University of Utah (UUMC), Primary Children's Medical Center (PCMC) and Intermountain Medical Center's (IMC) Neonatal Intesive Care Unit (NICUs)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Serum cytokine content | 6 hrs
  Plasma samples will be analyzed for the protein content of 13 different cytokines via a multiplexed sandwich capture assay performed at the ARUP Institute for Experimental and Clinical Pathology. The cytokines and chemokines assayed will include: CD40 ligand, interferon-gamma, interleukin-10, interleukin-12, interleukin-13, interleukin-1-β, interleukin-2, interleukin-2-receptor, interleukin-4, interleukin-5, interleukin-6, IL-8, and Tumor Necrosis Factor-alpha. In addition, we will assay components of the complement pathway including: total hemolytic complement, C3a, C5a, and FAB fragments in the alternative complement pathway. Cytokine protein levels before and after transfusion will be compared to each other and to the PRBC sample cytokine content.

SECONDARY OUTCOMES:
Assessment of NET formation | 6 hrs
  PMNs will be isolated from the participant blood samples following removal of the plasma via positive immunoselection. They will then be stimulated in vitro with NET-inducing stimuli such as lipopolysaccharide or platelet-activating factor for 1 hour under standard conditions and assayed for NET formation both qualitatively via confocal microscopy and quantitatively via histone H3 supernatant content as determined by ELISA and/or western blotting.

OTHER OUTCOMES:
Tissue oxygenation indexes (TOI) of cerebral (TOI brain ) and splanchnic (TOIabdo) regions | 53 hrs
  Tissue oxygenation indexes (TOI) of cerebral (TOI brain ) and splanchnic (TOIabdo) regions will be measured using NIRS and the values reported as CSOR (TOIabdo/TOI brain). Measurements will be continuously recorded and data points obtained for 30 minute periods at baseline or T0 (prior to PRBC transfusion), and every hour during the RBC transfusion (T1, T2, T3 and T4)
Mesenteric rSO2 | 53 hrs
  To determine whether alterations in mesenteric rSO2 can predict the development of NEC in VLBW infants.
  For this aim, TOI and CSOR will be measured every 3 hours for 30 minute periods in the first 48 hours following RBC transfusion (T5 to T16)(Table 1). By obtaining measurements during this time frame, we intend to capture the period of greatest susceptibility to develop NEC in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wiedmeier, MD, Principal Investigator — University of Utah; Mariana Baserga, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah

REFERENCES:
- [Background] Horbar JD, Badger GJ, Carpenter JH, Fanaroff AA, Kilpatrick S, LaCorte M, Phibbs R, Soll RF; Members of the Vermont Oxford Network. Trends in mortality and morbidity for very low birth weight infants, 1991-1999. Pediatrics. 2002 Jul;110(1 Pt 1):143-51. doi: 10.1542/peds.110.1.143. PMID 12093960
- [Background] Lemons JA, Bauer CR, Oh W, Korones SB, Papile LA, Stoll BJ, Verter J, Temprosa M, Wright LL, Ehrenkranz RA, Fanaroff AA, Stark A, Carlo W, Tyson JE, Donovan EF, Shankaran S, Stevenson DK. Very low birth weight outcomes of the National Institute of Child health and human development neonatal research network, January 1995 through December 1996. NICHD Neonatal Research Network. Pediatrics. 2001 Jan;107(1):E1. doi: 10.1542/peds.107.1.e1. PMID 11134465
- [Background] Stoll BJ. Epidemiology of necrotizing enterocolitis. Clin Perinatol. 1994 Jun;21(2):205-18. doi: 10.1016/S0095-5108(18)30341-5. PMID 8070222
- [Background] Mally P, Golombek SG, Mishra R, Nigam S, Mohandas K, Depalhma H, LaGamma EF. Association of necrotizing enterocolitis with elective packed red blood cell transfusions in stable, growing, premature neonates. Am J Perinatol. 2006 Nov;23(8):451-8. doi: 10.1055/s-2006-951300. Epub 2006 Sep 28. PMID 17009195
- [Background] Christensen RD, Lambert DK, Henry E, Wiedmeier SE, Snow GL, Baer VL, Gerday E, Ilstrup S, Pysher TJ. Is "transfusion-associated necrotizing enterocolitis" an authentic pathogenic entity? Transfusion. 2010 May;50(5):1106-12. doi: 10.1111/j.1537-2995.2009.02542.x. Epub 2009 Dec 29. PMID 20051059
- [Background] Josephson CD, Wesolowski A, Bao G, Sola-Visner MC, Dudell G, Castillejo MI, Shaz BH, Easley KA, Hillyer CD, Maheshwari A. Do red cell transfusions increase the risk of necrotizing enterocolitis in premature infants? J Pediatr. 2010 Dec;157(6):972-978.e1-3. doi: 10.1016/j.jpeds.2010.05.054. Epub 2010 Jul 21. PMID 20650470
- [Background] Blau J, Calo JM, Dozor D, Sutton M, Alpan G, La Gamma EF. Transfusion-related acute gut injury: necrotizing enterocolitis in very low birth weight neonates after packed red blood cell transfusion. J Pediatr. 2011 Mar;158(3):403-9. doi: 10.1016/j.jpeds.2010.09.015. Epub 2010 Nov 10. PMID 21067771
- [Background] Singh R, Visintainer PF, Frantz ID 3rd, Shah BL, Meyer KM, Favila SA, Thomas MS, Kent DM. Association of necrotizing enterocolitis with anemia and packed red blood cell transfusions in preterm infants. J Perinatol. 2011 Mar;31(3):176-82. doi: 10.1038/jp.2010.145. Epub 2011 Jan 27. PMID 21273983
- [Background] El-Dib M, Narang S, Lee E, Massaro AN, Aly H. Red blood cell transfusion, feeding and necrotizing enterocolitis in preterm infants. J Perinatol. 2011 Mar;31(3):183-7. doi: 10.1038/jp.2010.157. Epub 2011 Jan 20. PMID 21252964